CLINICAL TRIAL: NCT05962645
Title: A Phase 1 Study to Confirm the Single- and Multiple-dose Pharmacokinetics and to Evaluate Food Effect of Vapendavir in Healthy Participants and Participants With COPD
Brief Title: Phase 1 Study Into Pharmacokinetics and Food Effect of Vapendavir in Healthy Participants and Participants With COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altesa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALT VPV-101
Record Dates: First submitted 2023-06-07; First posted 2023-07-27 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: COPD; Respiratory Disease; Lower Respiratory Disease; Pulmonary Disease; Healthy
Keywords: Placebo; Parallel; Interventional; Clinical trial; Clinical study; Placebo-Controlled; Phase 1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiration Disorders; Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Healthy Participants (HP)
  Interventions: Drug: Vapendavir
- Group B (Experimental): Participants with COPD
  Interventions: Drug: Vapendavir

INTERVENTIONS:
Drug: Vapendavir — This study will measure and compare how VPV is absorbed in the blood, broken down in the body and eliminated when two 250 mg VPV tablets (500mg) are given in three different ways: A single dose, once a day, under fasted conditions (without any food); twice a day, for 7 days; and a single dose, once a day under fed conditions, after consuming a high-fat meal.

SUMMARY:
Vapendavir (VPV) is potent virostatic antiviral agent active against all known enterovirus species. VPV binds to the viral capsid, thereby inhibiting viral attachment to the target cell and, independently, preventing release of viral RNA (ribonucleic acid) into the cell. Alt VPV-101 is meant to investigate vapendavir in patients with chronic obstructive pulmonary disease (COPD) who develop a rhinoviral infection. This is a Phase 1, open-label, unblinded study. The primary objective of this study is to characterize single and multiple dose (plus a loading dose) plasma PK profiles of VPV in healthy participants (Group A) and participants with COPD (Group B). Group A is an open-label, 2-sequence, and up to a 3-period, cross-over study to assess the single-dose PK parameters and safety of VPV. Healthy participants may opt to participate in only the first 2 periods, all 3 periods or BID dosing, but it is preferred that participants complete all 3 periods. Group B is an open-label, multi-dose investigation of VPV PK parameters and safety in participants with COPD. Post-dose, follow up will continue for a minimum of 14 days and a maximum of 30 days, depending on which Group the participant is in and which periods said participant completes. There is a target for up to 24 adult participants comprised of healthy participants and participants with COPD.

DETAILED DESCRIPTION:
Vapendavir (VPV) has been in development for the treatment of infections with human rhinovirus (RV) and other respiratory enteroviruses for over a decade, with over 640 healthy adults and participants with Asthma receiving treatment across 7 clinical studies. Vapendavir is a potent and broad spectrum virostatic agent active against > 97% of RV A and B serotypes (no available assay for RV C, but clinical data indicate sensitivity similar to A and B), and 89% of other enteroviruses evaluated. Vapendavir has exhibited an acceptable safety and tolerability profile, to date, with no appreciable safety concerns with single doses up to 1056 milligram (mg) and daily doses up to 528 mg (264 mg twice daily), for up to 6 or 10 days.

ELIGIBILITY:
Inclusion Criteria: Healthy Participants (Group A)

1. Male or female participants, ≥ 18 and ≤ 55 years of age.
2. Weight ≥ 45 kilograms (kg), females and ≥ 50 kilograms, males.
3. Body mass index (BMI) within 18 to 32 kg/m2.
4. Female participants of childbearing potential must have a negative pregnancy test and females of non-childbearing potential must be post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented FSH levels ≥ 40 mIU/mL or be surgically sterile (bilateral oophorectomy, bilateral salpingectomy, hysterectomy or tubal ligation) at least 3 months prior to dosing.
5. If sexually active and/or of child-bearing potential (both females and males), must agree to abstinence or to use a highly effective forms of contraception ≥ 28 days prior to the first dose (females), during the study period (both males and females) and for 30 days (females) or 90 days (males) after the last dose.

   Examples: female participants: non-hormonal intrauterine device, double barrier; males (including those with a vasectomy): agree to use a condom and if a female partner of childbearing potential, use of at least one other contraceptive method; males must also agree not to donate sperm within 90 days after the last dose.

   Note: Refer to Section 12.5 for acceptable forms of contraception and timing required.
6. If participant becomes pregnant during the study or follow-up period, they agree to transmit all relevant safety information regarding the pregnancy and outcomes to the Sponsor or their designee (female partners of male participants will be asked to consent to the same), as requested.
7. Participants must be willing and able to understand and provide written informed consent.
8. Participants who are able and willing to adhere to the study visit schedule and other protocol requirements.

Inclusion Criteria: Participants with COPD (Group B)

1. ≥ 40 and ≤ 75 years of age.
2. BMI within 18 to 40 kg/m2.
3. Documented diagnosis of clinically stable COPD (no exacerbations within 45 days prior to study-drug administration), consistent with one these GOLD categories:

   • GOLD A: Minimally symptomatic, low risk of future exacerbations (ie, mMRC grade 0 to 1 or CAT score < 10; 0 to 1 exacerbation per year and no prior hospitalization for exacerbation).

   • GOLD B: More symptomatic, low risk of future exacerbations (ie, mMRC grade ≥ 2 or CAT score ≥ 10; 0 to 1 exacerbation per year and no prior hospitalization for exacerbation).

   • GOLD C: Minimally symptomatic, high risk of future exacerbations (ie, mMRC grade 0 to 1 or CAT score < 10; ≥ 2 exacerbations per year or ≥ 1 hospitalization for exacerbation).
4. Must be taking as directed, at least one medication for the management of COPD. For GOLD A patients, medication could be for use only as needed. GOLD B and C patients should be on at least one active chronic therapy, consistent with treatment guidelines.
5. Female participants of childbearing potential must have a negative pregnancy test and females of non-childbearing potential must be post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented FSH levels ≥ 40 mIU/mL or be surgically sterile (bilateral oophorectomy, bilateral salpingectomy, hysterectomy or tubal ligation) at least 3 months prior to dosing.
6. If sexually active and/or of child-bearing potential (both females and males), must agree to abstinence or to use a highly effective forms of contraception ≥ 28 days prior to the first dose (females), during the study period (both males and females) and for 30 days (females) or 90 days (males) after the last dose.

   Examples: female participants: non-hormonal intrauterine device, double barrier; males (including those with a vasectomy): agree to use a condom and if a female partner of childbearing potential, use of at least one other contraceptive method; males must also agree not to donate sperm within 90 days after the last dose.
7. If participant becomes pregnant during the study or follow-up period, they agree to transmit all relevant safety information regarding the pregnancy and outcomes to the Sponsor or their designee (female partners of male participants will be asked to consent to the same), as requested.
8. Participants must be willing and able to understand and provide written informed consent.
9. Participants who are able and willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria: Healthy Participants (Group A)

1. Any clinically significant illness and/or surgery within 4 weeks prior to dosing. This includes but is not limited to uncontrolled and clinically significant neurologic (including seizure disorders), cardiovascular, central nervous system (CNS), pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic (including allergic skin rash), hematologic or endocrine disease, psychiatric disorder or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
2. Any clinically significant finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking VPV, or a similar drug in the same class, or that might interfere with the conduct of the study.

   Note: It is the responsibility of the Investigator to assess the clinical significance of medical history or ongoing findings; however, consultation with the Medical Monitor may be warranted.
3. The participant has current or recent (within 28 days) gastrointestinal disease significant enough in the opinion of the Investigator that it would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn), or any clinically significant gastric surgical intervention that could impact study drug absorption characteristics, in the opinion of the Investigator.
4. History or current condition where repeat blood draws pose more than minimal risk to participant (eg, hemophilia, other severe coagulation disorders).
5. Significantly impaired venous access and/or inability to tolerate repeat blood draws.
6. Use of nicotine-containing products (including but not limited to electronic cigarettes, cigarettes, pipes, cigars, chewing tobacco, snuff, nicotine patch or gum) within 10 h of 1st dose in a Period, and within 2h (± 30 minutes) of any other dose, and unwillingness to adhere to requirements for duration of study.
7. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
8. Positive drug or alcohol test at the screening.
9. Pregnant (documented test) or nursing female participants at screening.
10. Sexually active participants/female partner(s) of childbearing potential who are unwilling to utilize protocol-defined acceptable forms of contraception for duration of study and follow-up period.
11. Participants using hormonal contraceptives and/or estrogen-based hormone replacement therapy via any route ≤ 14 days prior to dosing.
12. Donation or loss of ≥ 450 mL of participant's blood volume (including plasmapheresis) or transfusion of any blood product within 45 days prior to first dose of study drug and agree not to donate for 45 days after completion of the study.
13. Any clinically significant ECG abnormalities, including QT interval with Fridericia correction method (QTcF) ≥ 450 msec (males) or ≥ 470 msec (females) or PR interval outside the range of 120 to 220 msec, confirmed with1 repeat testing, at screening.
14. A seated or semi-supine blood pressure outside of the range of 85 to 145 mm Hg for systolic and 50 to 95 mm Hg for diastolic confirmed on repeat testing within a maximum of 30 minutes, at screening.
15. A resting heart rate outside of the range of 40 to 100 beats per minute, confirmed on repeat testing within a maximum of 30 minutes, at screening.
16. Any dietary restrictions or preferences that may interfere with the conduct of the study.
17. The participant has a history of suicidal ideation/behavior within 6 years or presents with such at screening.
18. The participant has a positive test result for: hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody without evidence of curative treatment, or human immunodeficiency virus (HIV) antibody/antigen at Screening or a known history of HIV infection.
19. Participation in another clinical study with an investigational agent within 30 days for small molecules, 90 days for biologics, or 5 half-lives (whichever is longer) of planned baseline and during study.
20. Renal impairment (eg, estimated glomerular filtration rate (eGFR) calculated using CKD- EPI 2021 equation, limit < 60) (17, 18).
21. Hepatic disease (clinically significant abnormal liver function laboratory test results (eg, ALT, AST, gamma glutamyl transferase (GGT), alkaline phosphatase (ALP), total bilirubin ≥ 1.5 the upper limit of normal).
22. Use of medications/agents ≤ 28 days of baseline and during study that may alter clearance by CYP3A4 or 2C19 (eg, strong inhibitors or inducers); see Table 7 for reference.
23. Prescription or over-the-counter (OTC) medications and natural health products (including but not limited to herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements) that cannot be safely discontinued within 7 days prior to dosing (14 days if a potential other enzyme inhibitor/inducer), or up to 5 half-lives (whichever is longer), with the exception of the occasional use (up to 2 g daily) of acetaminophen.
24. Any vaccine, including COVID-19 vaccine, within 14 days prior to dosing.
25. Depot injection or implant of any drug for 3 months prior to dosing.
26. Consumption of grapefruit or grapefruit juice or grapefruit-related citrus fruits (eg, Seville oranges, pomelos) within the 7 days prior to planned Study baseline and during study.
27. A condition that requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being.
28. Known allergic reaction to vapendavir, related drug classes, or to any excipients in the formulation.
29. History of illicit drug abuse and/or use within 3 months prior to screening; "soft" drugs (eg, tetrahydrocannabinol-containing agents, which may be legal in some settings) are prohibited within 28 days of dosing.
30. In the opinion of the Principal Investigator (PI), other findings (eg, unexplained clinically significant screening lab abnormalities, physical/psychologic issues), that would make the participant unsuitable for study participation.

Exclusion Criteria: Participants with COPD (Group B)

1. Exacerbation of COPD within 45 days prior to study-drug administration.
2. Use of nicotine-containing products (including but not limited to electronic cigarettes, cigarettes, pipes, cigars, chewing tobacco, snuff, nicotine patch or gum) within 10 h of 1st dose in a Period, and within 2h (± 30 minutes) of any other dose, and unwillingness to adhere to requirements for duration of study.
3. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
4. Positive drug or alcohol test at the screening.
5. Pregnant (documented test) or nursing female participants at screening.
6. Sexually active participants/female partner(s) of childbearing potential who are unwilling to utilize protocol-defined acceptable forms of contraception for duration of study and follow-up period.
7. Participants using hormonal contraceptives and/or estrogen-based hormone replacement therapy via any route ≤ 14 days prior to dosing.
8. Donation or loss of ≥ 450 mL of participant's blood volume (including plasmapheresis) or transfusion of any blood product within 45 days prior to first dose of study drug and agree not to donate for 45 days after completion of the study.
9. Any clinically significant ECG abnormalities, including QT interval with Fridericia correction method (QTcF) ≥ 450 msec (males) or ≥ 470 msec (females) or PR interval outside the range of 120 to 220 msec, confirmed with1 repeat testing, at screening.
10. A seated or semi-supine blood pressure outside of the range of 85 to 145 mm Hg for systolic and 50 to 95 mm Hg for diastolic confirmed on repeat testing within a maximum of 30 minutes, at screening.
11. A resting heart rate outside of the range of 40 to 100 beats per minute, confirmed on repeat testing within a maximum of 30 minutes, at screening.
12. Any dietary restrictions or preferences that may interfere with the conduct of the study.
13. The participant has a history of suicidal ideation/behavior within 6 years or presents with such at screening.
14. The participant has a positive test result for: hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody without evidence of curative treatment, or human immunodeficiency virus (HIV) antibody/antigen at Screening or a known history of HIV infection.
15. Any unstable clinically significant finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking VPV, or a similar drug in the same class, or that might interfere with the conduct of the study.

    Note: It is the responsibility of the Investigator to assess the clinical significance and stability of conditions noted in the medical history and of ongoing findings; however, consultation with the Medical Monitor may be warranted.
16. The participant has current or recent (within 28 days) gastrointestinal disease significant enough in the opinion of the Investigator that it would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn), or any clinically significant gastric surgical intervention that could impact study drug absorption characteristics, in the opinion of the Investigator.
17. History or current condition where repeat blood draws pose more than minimal risk to participant (eg, hemophilia, other severe coagulation disorders).
18. Significantly impaired venous access and/or inability to tolerate repeat blood draws.
19. Diagnosed with Type 1 diabetes, controlled or otherwise.
20. Renal impairment (eg, estimated glomerular filtration rate (eGFR) calculated using CKD- EPI 2021 equation, limit < 60) (17, 18).
21. Hepatic disease (clinically significant abnormal liver function laboratory test results (eg, ALT, AST, gamma glutamyl transferase (GGT), alkaline phosphatase (ALP), total bilirubin ≥ 1.5 the upper limit of normal).
22. Uncontrolled comorbid conditions, as defined below:

    * Other than COPD, other ongoing chronic medical diagnoses or conditions (eg, hypertension, hypercholesteremia, Type 2 diabetes, osteoarthritis), except those excluded as noted above, must be controlled, which is defined as stable for the last 90 days (no hospitalizations, emergency room (ER) or urgent care for condition (excluding musculoskeletal conditions).
    * Subjects may be on relevant medications for the controlled conditions noted above only if:

1. The condition or disease for which they're prescribed is stable and not deteriorating, 2. Medications to manage the stable comorbid conditions (including prescription or OTC medications and natural health products (including but not limited to herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements)) are not otherwise listed as excluded in the exclusion criteria (eg, drugs of abuse, those that inhibit/induce CYP3A4 or 2C19 noted in Table 7), and, 3. Medications pose no additional risk to subject safety, assessment of adverse events or pharmacokinetics.

* This also includes no change in prescription medication, dose or frequency resulting from new symptoms or deterioration of the medical diagnosis or condition in the 90 days prior to enrollment (note: restrictions includes changes in routine/as needed (PRN) use).
* Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, so long as in the same class of medication, will not be considered a deviation of this criterion.
* Any change in prescription medication due to improvement of a disease outcome (eg, lowering of the dosage or frequency), as determined by the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572, will not be considered a deviation of this inclusion criterion.

  23. Use of medications/agents ≤ 28 days of baseline and during study that may alter clearance by CYP3A4 or 2C19 (eg, strong inhibitors or inducers); see Table 7 for reference.

  24. Any vaccine, including COVID-19 vaccine, within 14 days prior to dosing. 25. Depot injection or implant of any drug for 3 months prior to dosing. 26. Consumption of grapefruit or grapefruit juice or grapefruit-related citrus fruits (eg, Seville oranges, pomelos) within the 7 days prior to planned study baseline and during study.

  27. Known allergic reaction to vapendavir, related drug classes, or to any excipients in the formulation.

  28. History of illicit drug abuse and/or use within 3 months prior to screening; "soft" drugs (eg, tetrahydrocannabinol-containing agents, which may be legal in some settings) are prohibited within 28 days of dosing.

  29. In the opinion of the PI, other findings (eg, unexplained clinically significant screening lab abnormalities, physical/psychologic issues), that would make the participant unsuitable for study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Analyses | Through study completion, up to 3 weeks
  Plasma PK parameters for each participant will be estimated from the plasma concentrations of VPV over the sampling interval using standard non-compartmental PK analysis method. Additional PK parameters may be analyzed as appropriate.
  PK parameters will be summarized by group, treatment, period, and study day using descriptive statistics.
  Food effect on single-dose PK of VPV will be evaluated with fasted/fed status as a fixed effect and participant as a random effect.
  VPV Peak Plasma Concentration (Cmax)
  There will also be exploratory descriptive comparisons on PK parameters to explore any potential differences (e.g., healthy participants relative to participants with COPD, concomitant medication use, BMI, age).
Pharmacokinetic Analyses | Through study completion, up to 3 weeks
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: David Wyatt, MD, Principal Investigator — VP Medical Affairs
Locations (1):
- Syneos Health Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The Sponsor or their designee will be responsible for generating a final clinical study report.
  Final study results will be shared with regulatory authorities and may also be posted on Clincaltrials.gov or other publicly accessible sites, as required.
  All data generated from this study shall be held in strict confidence along with all information furnished by the Sponsor. The Sponsor acknowledges the importance of public disclosure/ publication of information collected or generated by the Institution and Principal Investigator. However, independent analyses and/or publication of these data by the Investigator or any member of his/her staff are not permitted without prior written consent of the Sponsor.

REFERENCES:
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Kaiser L, Crump CE, Hayden FG. In vitro activity of pleconaril and AG7088 against selected serotypes and clinical isolates of human rhinoviruses. Antiviral Res. 2000 Sep;47(3):215-20. doi: 10.1016/s0166-3542(00)00106-6. PMID 10974374
- [Background] Barnard DL, Hubbard VD, Smee DF, Sidwell RW, Watson KG, Tucker SP, Reece PA. In vitro activity of expanded-spectrum pyridazinyl oxime ethers related to pirodavir: novel capsid-binding inhibitors with potent antipicornavirus activity. Antimicrob Agents Chemother. 2004 May;48(5):1766-72. doi: 10.1128/AAC.48.5.1766-1772.2004. PMID 15105133
- [Background] Sykes A, Johnston SL. Etiology of asthma exacerbations. J Allergy Clin Immunol. 2008 Oct;122(4):685-688. doi: 10.1016/j.jaci.2008.08.017. PMID 19014758
- [Background] Hayden FG. Rhinovirus and the lower respiratory tract. Rev Med Virol. 2004 Jan-Feb;14(1):17-31. doi: 10.1002/rmv.406. PMID 14716689
- [Background] Newcomb DC, Peebles RS Jr. Bugs and asthma: a different disease? Proc Am Thorac Soc. 2009 May 1;6(3):266-71. doi: 10.1513/pats.200806-056RM. PMID 19387028
- [Background] Mallia P, Message SD, Kebadze T, Parker HL, Kon OM, Johnston SL. An experimental model of rhinovirus induced chronic obstructive pulmonary disease exacerbations: a pilot study. Respir Res. 2006 Sep 6;7(1):116. doi: 10.1186/1465-9921-7-116. PMID 16956406
- [Background] Message SD, Laza-Stanca V, Mallia P, Parker HL, Zhu J, Kebadze T, Contoli M, Sanderson G, Kon OM, Papi A, Jeffery PK, Stanciu LA, Johnston SL. Rhinovirus-induced lower respiratory illness is increased in asthma and related to virus load and Th1/2 cytokine and IL-10 production. Proc Natl Acad Sci U S A. 2008 Sep 9;105(36):13562-7. doi: 10.1073/pnas.0804181105. Epub 2008 Sep 3. PMID 18768794
- [Background] Wheaton AG, Cunningham TJ, Ford ES, Croft JB; Centers for Disease Control and Prevention (CDC). Employment and activity limitations among adults with chronic obstructive pulmonary disease--United States, 2013. MMWR Morb Mortal Wkly Rep. 2015 Mar 27;64(11):289-95. PMID 25811677
- [Background] Zafari Z, Li S, Eakin MN, Bellanger M, Reed RM. Projecting Long-term Health and Economic Burden of COPD in the United States. Chest. 2021 Apr;159(4):1400-1410. doi: 10.1016/j.chest.2020.09.255. Epub 2020 Oct 2. PMID 33011203
- [Background] Halpin DMG, Criner GJ, Papi A, Singh D, Anzueto A, Martinez FJ, Agusti AA, Vogelmeier CF. Global Initiative for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease. The 2020 GOLD Science Committee Report on COVID-19 and Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2021 Jan 1;203(1):24-36. doi: 10.1164/rccm.202009-3533SO. PMID 33146552
- [Background] Altesa Biosciences Inc. Investigator's Brochure for Vapendavir v 10. 2023
- [Background] Abzug MJ, Michaels MG, Wald E, Jacobs RF, Romero JR, Sanchez PJ, Wilson G, Krogstad P, Storch GA, Lawrence R, Shelton M, Palmer A, Robinson J, Dennehy P, Sood SK, Cloud G, Jester P, Acosta EP, Whitley R, Kimberlin D; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. A Randomized, Double-Blind, Placebo-Controlled Trial of Pleconaril for the Treatment of Neonates With Enterovirus Sepsis. J Pediatric Infect Dis Soc. 2016 Mar;5(1):53-62. doi: 10.1093/jpids/piv015. Epub 2015 Apr 16. PMID 26407253
- [Background] US Food and Drug Administration Center for Drug Evaluation and Research. Draft Guidance: Assessing the Effects of Food on Drugs in INDs and NDAs - Clinical Pharmacology Considerations Guidance for Industry. 2019.
- [Background] Proud D. Host response to human rhinovirus infection: toward targeted treatment strategies. Future Virology 2009; 4: 97-10
- See also: Sponsor website — https://altesabio.com/